CLINICAL TRIAL: NCT00212303
Title: Exercise Training in Type 2 Diabetes and Hypertension
Acronym: SHAPE2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kerry Stewart, Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK62368 (completed); DK62368
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes; Hypertension
Keywords: type 2 diabetes; hypertension; exercise training; cardiac, peripheral; body composition; physical fitness; inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise training (Experimental): Exercise training, 3 times per week, for 6 months.
  Interventions: Behavioral: Exercise training for 6 months
- Control (No Intervention): Usual care no active exercise intervention

INTERVENTIONS:
Behavioral: Exercise training for 6 months — Exercise 3 times/week for 6 months. Exercise consists of aerobic and resistance exercise
  Arms: Exercise training

SUMMARY:
The coexistence of diabetes and hypertension is damaging to cardiac and peripheral vascular structure and function. Although several health organizations endorse exercise training as a treatment for type 2 diabetes, most studies of exercise and diabetes have focused on controlling blood sugar but not on cardiovascular health. The aim of this study is to determine if exercise training reduces blood pressure and improves cardiovascular health in persons who have both type 2 diabetes and hypertension. An equal number of men and women will be enrolled, and another aim of the study is to examine gender differences in response to exercise training.

DETAILED DESCRIPTION:
Type 2 diabetes is associated with damage, dysfunction, and failure of various organs. The coexistence of diabetes and hypertension is particularly damaging to cardiac and peripheral vascular structure and function. These diseases, either alone or combined, result in increased left ventricular mass and wall thickness, left ventricular diastolic dysfunction, impaired endothelial vasodilator function, and increased vascular stiffness. Although several health organizations endorse exercise training as a therapeutic modality for type 2 diabetes, most studies of exercise and diabetes have focused on glycemic control but not on cardiovascular health. Although exercise lowers blood pressure in persons without diabetes, there are profound gaps in knowledge about the effects of exercise training on blood pressure and cardiovascular health in persons with type 2 diabetes. The primary specific aim of this study is to determine if exercise training reduces blood pressure in persons who have both type 2 diabetes and high normal blood pressure or mild hypertension prehypertension or Stage 1 (mild) hypertension. Subjects will be randomized to 6-months of exercise training, consistent with established guidelines for diabetes and for hypertension, or to a usual care control group. The second specific aim is to identify the effects of exercise training on parameters of cardiac and peripheral vascular structure and function related to cardiovascular disease in diabetes and hypertension. We will assess left ventricular mass, left ventricular diastolic function, endothelial vasodilator function, and vascular stiffness using high-resolution ultrasound, Doppler echocardiography, and magnetic resonance imaging. We will also examine interleukin-6 and high-resolution C-reactive protein as novel risk factors for cardiovascular disease and diabetes to determine the effects of exercise training on the inflammatory process. Because exercise training improves fitness and may improve body composition and regional fat distribution, the associations of change in these parameters with change in blood pressure and cardiac and peripheral vascular structure and function will be analyzed. An equal number of men and women will be enrolled, and a third specific aim of the study is to examine gender differences in response to exercise training. This study will expand the scientific knowledge that defines exercise guidelines and will provide new insight into the mechanisms by which exercise reduces blood pressure and improves cardiovascular health in persons with type 2 diabetes and hypertension.

ELIGIBILITY:
Inclusion Criteria:

ages 40-65 years type 2 diabetes BP between SBP 120-159 or DBP 80-99 mm Hg sedentary

Exclusion Criteria:

cardiovascular disease abnormal exercise stress test smoking insulin use major illnesses that would preclude exercise training pregnancy in women engaged in regular exercise or weight loss diet program substance abuse morbid obesity BMI > 42

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2004-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure at 6 months | 6 months

SECONDARY OUTCOMES:
Cardiac and peripheral structure and function at 6 months | 6 months
Fitness and body composition at 6 months | 6 months
Cardiac and diabetes risk factors at 6 months | 6 months
Systemic inflammation at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerry J Stewart, EdD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Dobrosielski DA, Barone Gibbs B, Chaudhari S, Ouyang P, Silber HA, Stewart KJ. Effect of exercise on abdominal fat loss in men and women with and without type 2 diabetes. BMJ Open. 2013 Nov 25;3(11):e003897. doi: 10.1136/bmjopen-2013-003897. PMID 24282247
- [Derived] Barone Gibbs B, Dobrosielski DA, Althouse AD, Stewart KJ. The effect of exercise training on ankle-brachial index in type 2 diabetes. Atherosclerosis. 2013 Sep;230(1):125-30. doi: 10.1016/j.atherosclerosis.2013.07.002. Epub 2013 Jul 14. PMID 23958264
- [Derived] Nam S, Dobrosielski DA, Stewart KJ. Predictors of exercise intervention dropout in sedentary individuals with type 2 diabetes. J Cardiopulm Rehabil Prev. 2012 Nov-Dec;32(6):370-8. doi: 10.1097/HCR.0b013e31826be485. PMID 23011489
- [Derived] Gibbs BB, Dobrosielski DA, Lima M, Bonekamp S, Stewart KJ, Clark JM. The association of arterial shear and flow-mediated dilation in diabetes. Vasc Med. 2011 Aug;16(4):267-74. doi: 10.1177/1358863X11411361. Epub 2011 Jun 27. PMID 21708874
- [Derived] Moseley KF, Dobrosielski DA, Stewart KJ, Sellmeyer DE, Jan De Beur SM. Lean mass predicts hip geometry in men and women with non-insulin-requiring type 2 diabetes mellitus. J Clin Densitom. 2011 Jul-Sep;14(3):332-9. doi: 10.1016/j.jocd.2011.04.007. Epub 2011 Jun 11. PMID 21652249
- [Derived] Bennett WL, Ouyang P, Wu AW, Barone BB, Stewart KJ. Fatness and fitness: how do they influence health-related quality of life in type 2 diabetes mellitus? Health Qual Life Outcomes. 2008 Dec 4;6:110. doi: 10.1186/1477-7525-6-110. PMID 19055828